CLINICAL TRIAL: NCT05958641
Title: Early Warning Model Construction on Cognition, Resistance and Using Risk of the New Psychoactive Substances in Adolescents Based on Behavioral Expression of Addiction Susceptibility Genes and Adverse Childhood Experience
Brief Title: Construction of Early Warning Model for the New Psychoactive Substances Using in Adolescents
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wei XIA, PhD (Other)
Responsible Party: Sponsor-Investigator, Wei XIA, PhD, Associate Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: 202310893
Record Dates: First submitted 2023-07-16; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Drug Addiction
Keywords: risk prediction model; NPS; addiction susceptibility genes; adverse childhood experience; adolescents
MeSH Terms: conditions — Substance-Related Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Investigation Team: Questionnaires assessed adolescents aged 14-35 years old (including 14,25 years old) who agreed to participate in the study
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Participants will be asked to complete the questionnaire including general demographic information, the cognition, resistance and use of NPS as well as the behavioral expression of addiction susceptibility genes and adverse childhood experience.

SUMMARY:
Based on the biological-psychology-sociological medicine pattern, this study aims to construction an early warning model of the New Psychoactive Substances (NPS) using for adolescents aged 14-35 years old. This study intends to obtain the data related to the behavioral expression of addiction susceptibility genes, adverse childhood experience, cognition, resistance and the use of NPS in adolescents by questionnaire survey (sample size: 200), and then use logistic regression and machine learning to construct an early warning model.

DETAILED DESCRIPTION:
Based on the biological-psychology-sociological medicine pattern, this study aims to construction an early warning model on the use of the New Psychoactive Substances using for adolescents aged 14-35 years old. This study intends to conduct a questionnaire survey (sample size 200) to obtain data related to the behavioral expression of addiction susceptibility genes, childhood adversity experience, cognition, resistance and the use of NPS in adolescents from different regions and different populations. Through data analysis, this study aims to get the weight of different risk factors on NPS use, and then use logistic regression and machine learning to construct an early warning model, so as to screen out high-risk groups. At the same time, the expert group was consulted to establish a risk early warning system to provide a basis for intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 14-35 (including 14,35 years old)
* Agree to participate in the studies

Exclusion Criteria:

* Be diagnosed with psychological or mental illness
* People that are unconscious, emotionally unstable, or unable to communicate normally
* Patients with severe diseases

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: General adolescents between 14-35 years old
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-17 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
the cognition of NPS | Baseline
  knowledge questionnaire of drug types and risk awareness of drug use will be investigated to know the degree of cognition to NPS
the resistance of NPS | Baseline
  the drug refusal self-efficacy scale and the drug use permissive attitude will be used to measure the the resistance of NPS
the use of NPS | Baseline
  there will be some questions to investigate the drug use conditions
Adverse Childhood Experience | Baseline
  the Chinese version of Adverse Childhood Experience Scale with 10 items will be used to measure the adverse childhood experience
hedonic hunger | Baseline
  the Power of Food Scale with 15 items will be used to measure hedonic hunger
sensation seeking personality | Baseline
  the Brief Sensation Seeking Scale for Chinese with 8 items will be used to measure sensation seeking personality
prosocial behavior | Baseline
  the Prosocial Tendencies Measure with 26 items will be used to measure prosocial behavior
externalizing behavior | Baseline
  17 items of aggressive behavior and 15 items of rule-breaking behavior from the Chinese Version of Achenbach Youth Self-Report-2001 Version will be used to measure adolescents' degree of externalizing behavior
sleep quality | Baseline
  the Pittsburgh Sleep Quality Index with 9 items will be used to measure adolescents' sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No